CLINICAL TRIAL: NCT05611866
Title: A Pilot Study of Fecal Microbiota Transplant (FMT) and Its Effects in Patients With Crohn's Disease With Moderate-to-High Risk of Colonization of Adherent-Invasive E. Coli (AIEC)
Brief Title: A Pilot Study of FMT on CD Patients With AIEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT CD AIEC study
Record Dates: First submitted 2022-10-14; First posted 2022-11-10 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Crohn Disease
Keywords: Fecal Microbiota Transplant; Adherent-invasive Escherichia coli
MeSH Terms: conditions — Crohn Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: All recruited patients will receive FMT.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): Recruited patients will receive Fecal Microbiota Transplantation
  Interventions: Procedure: Fecal Microbiota Transplantation

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — FMT at Week 0

SUMMARY:
The goal of this pilot study is to test whether Fecal Microbiota Transplant (FMT) would be an effective antibacterial treatment for managing Adherent-invasive Escherichia coli (AIEC) colonization in Crohn's disease (CD) patients.

It aims to assess the safety of FMT in patients with clinically inactive or mild to moderate CD and to determine the presence of AIEC before and after FMT.

Participants will receive FMT via colonoscopy and have a follow-up colonoscopy at the end of the study.

DETAILED DESCRIPTION:
Experimental and observational data suggest that intestinal inflammation in Crohn's Disease (CD) arises from abnormal immune response to intestinal microbiota in genetically susceptible individuals. Genes that regulate innate immune response, intestinal barrier function and bacteria killing of intracellular pathogens have been associated with an increased risk for developing CD in Caucasian populations. The search for specific pathogens in CD has identified in the intestinal mucosa of patients several candidates. One with much supporting evidence is the adherent invasive Escherichia coli (AIEC). Since its discovery in 1998, several groups have reported a higher prevalence of AIEC in CD patients compared to healthy subjects and confirmed their pro-inflammatory potential. A growing body of work indicates that different host environments can select such AIEC pathobiont. AIEC colonization in mice leads to strong inflammatory responses in the gut suggesting that AIEC could play a role in CD immunopathogenesis.

Faecal microbiota transplantation (FMT) represents a clinically feasible way to restore the gut microbial ecology and has proven to be a breakthrough for the treatment of recurrent Clostridium difficile infection. Clinical trials are being conducted to evaluate its use for other conditions including inflammatory bowel disease, irritable bowel syndrome, diabetes mellitus, non-alcoholic steatohepatitis and hepatic encephalopathy. Efficacy of FMT on CD endoscopic lesions and AIEC colonization remains to be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age;
* Patients with CD history ≥ 3-month duration;
* Patients with no or mild-to-moderate symptoms defined as Harvey Bradshaw Index (HBI) < 16 ;
* Patients with positive total E.coli antibodies (AEcAb)

Exclusion Criteria:

* Pregnancy;
* New biological treatment or steroids use within 4 weeks;
* Current Colorectal tumor;
* Active gastrointestinal bleeding;
* Having ulcerative colitis;
* Having colectomy or partial colectomy (less than ileo-transverse colonic anastomosis);
* Having colonic or small bowel stoma;
* Active perianal lesions;
* Receiving antibiotics within 4 weeks;
* Presenting psychological or linguistic incapability to sign the informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | 12 weeks
  Occurrence of any adverse events

SECONDARY OUTCOMES:
Change in AIEC colonization | Week 12
  Presence of mucosa-associated AIEC before and after receiving FMT
Change in inflammatory biomarker Erythrocyte sedimentation rate (ESR) | Week 12
Change in inflammatory biomarker C-reactive protein (CRP) | Week 12
Change in fecal microbiota | Week 12
  Fecal microbiota, including diversity, composition and functional capacity will be measured before and after receiving FMT
Disease Severity | Week 12
  Harvey Bradshaw Index score will be used to measure disease severity where scores higher than 16 indicate disease activity is severe

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan GG. The global burden of IBD: from 2015 to 2025. Nat Rev Gastroenterol Hepatol. 2015 Dec;12(12):720-7. doi: 10.1038/nrgastro.2015.150. Epub 2015 Sep 1. PMID 26323879
- [Background] Ng SC, Tang W, Ching JY, Wong M, Chow CM, Hui AJ, Wong TC, Leung VK, Tsang SW, Yu HH, Li MF, Ng KK, Kamm MA, Studd C, Bell S, Leong R, de Silva HJ, Kasturiratne A, Mufeena MNF, Ling KL, Ooi CJ, Tan PS, Ong D, Goh KL, Hilmi I, Pisespongsa P, Manatsathit S, Rerknimitr R, Aniwan S, Wang YF, Ouyang Q, Zeng Z, Zhu Z, Chen MH, Hu PJ, Wu K, Wang X, Simadibrata M, Abdullah M, Wu JC, Sung JJY, Chan FKL; Asia-Pacific Crohn's and Colitis Epidemiologic Study (ACCESS) Study Group. Incidence and phenotype of inflammatory bowel disease based on results from the Asia-pacific Crohn's and colitis epidemiology study. Gastroenterology. 2013 Jul;145(1):158-165.e2. doi: 10.1053/j.gastro.2013.04.007. Epub 2013 Apr 9. PMID 23583432
- [Background] Ng SC, Tang W, Leong RW, Chen M, Ko Y, Studd C, Niewiadomski O, Bell S, Kamm MA, de Silva HJ, Kasturiratne A, Senanayake YU, Ooi CJ, Ling KL, Ong D, Goh KL, Hilmi I, Ouyang Q, Wang YF, Hu P, Zhu Z, Zeng Z, Wu K, Wang X, Xia B, Li J, Pisespongsa P, Manatsathit S, Aniwan S, Simadibrata M, Abdullah M, Tsang SW, Wong TC, Hui AJ, Chow CM, Yu HH, Li MF, Ng KK, Ching J, Wu JC, Chan FK, Sung JJ; Asia-Pacific Crohn's and Colitis Epidemiology Study ACCESS Group. Environmental risk factors in inflammatory bowel disease: a population-based case-control study in Asia-Pacific. Gut. 2015 Jul;64(7):1063-71. doi: 10.1136/gutjnl-2014-307410. Epub 2014 Sep 12. PMID 25217388
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Jostins L, Ripke S, Weersma RK, Duerr RH, McGovern DP, Hui KY, Lee JC, Schumm LP, Sharma Y, Anderson CA, Essers J, Mitrovic M, Ning K, Cleynen I, Theatre E, Spain SL, Raychaudhuri S, Goyette P, Wei Z, Abraham C, Achkar JP, Ahmad T, Amininejad L, Ananthakrishnan AN, Andersen V, Andrews JM, Baidoo L, Balschun T, Bampton PA, Bitton A, Boucher G, Brand S, Buning C, Cohain A, Cichon S, D'Amato M, De Jong D, Devaney KL, Dubinsky M, Edwards C, Ellinghaus D, Ferguson LR, Franchimont D, Fransen K, Gearry R, Georges M, Gieger C, Glas J, Haritunians T, Hart A, Hawkey C, Hedl M, Hu X, Karlsen TH, Kupcinskas L, Kugathasan S, Latiano A, Laukens D, Lawrance IC, Lees CW, Louis E, Mahy G, Mansfield J, Morgan AR, Mowat C, Newman W, Palmieri O, Ponsioen CY, Potocnik U, Prescott NJ, Regueiro M, Rotter JI, Russell RK, Sanderson JD, Sans M, Satsangi J, Schreiber S, Simms LA, Sventoraityte J, Targan SR, Taylor KD, Tremelling M, Verspaget HW, De Vos M, Wijmenga C, Wilson DC, Winkelmann J, Xavier RJ, Zeissig S, Zhang B, Zhang CK, Zhao H; International IBD Genetics Consortium (IIBDGC); Silverberg MS, Annese V, Hakonarson H, Brant SR, Radford-Smith G, Mathew CG, Rioux JD, Schadt EE, Daly MJ, Franke A, Parkes M, Vermeire S, Barrett JC, Cho JH. Host-microbe interactions have shaped the genetic architecture of inflammatory bowel disease. Nature. 2012 Nov 1;491(7422):119-24. doi: 10.1038/nature11582. PMID 23128233
- [Background] Darfeuille-Michaud A, Boudeau J, Bulois P, Neut C, Glasser AL, Barnich N, Bringer MA, Swidsinski A, Beaugerie L, Colombel JF. High prevalence of adherent-invasive Escherichia coli associated with ileal mucosa in Crohn's disease. Gastroenterology. 2004 Aug;127(2):412-21. doi: 10.1053/j.gastro.2004.04.061. PMID 15300573
- [Background] Martinez-Medina M, Aldeguer X, Lopez-Siles M, Gonzalez-Huix F, Lopez-Oliu C, Dahbi G, Blanco JE, Blanco J, Garcia-Gil LJ, Darfeuille-Michaud A. Molecular diversity of Escherichia coli in the human gut: new ecological evidence supporting the role of adherent-invasive E. coli (AIEC) in Crohn's disease. Inflamm Bowel Dis. 2009 Jun;15(6):872-82. doi: 10.1002/ibd.20860. PMID 19235912
- [Background] Small CL, Reid-Yu SA, McPhee JB, Coombes BK. Persistent infection with Crohn's disease-associated adherent-invasive Escherichia coli leads to chronic inflammation and intestinal fibrosis. Nat Commun. 2013;4:1957. doi: 10.1038/ncomms2957. PMID 23748852
- [Background] Hansen JJ, Sartor RB. Therapeutic Manipulation of the Microbiome in IBD: Current Results and Future Approaches. Curr Treat Options Gastroenterol. 2015 Mar;13(1):105-20. doi: 10.1007/s11938-014-0042-7. PMID 25595930
- [Background] Nicolas-Chanoine MH, Bertrand X, Madec JY. Escherichia coli ST131, an intriguing clonal group. Clin Microbiol Rev. 2014 Jul;27(3):543-74. doi: 10.1128/CMR.00125-13. PMID 24982321
- [Background] Lubbert C, Straube L, Stein C, Makarewicz O, Schubert S, Mossner J, Pletz MW, Rodloff AC. Colonization with extended-spectrum beta-lactamase-producing and carbapenemase-producing Enterobacteriaceae in international travelers returning to Germany. Int J Med Microbiol. 2015 Jan;305(1):148-56. doi: 10.1016/j.ijmm.2014.12.001. Epub 2014 Dec 9. PMID 25547265
- [Background] Broaders E, Gahan CG, Marchesi JR. Mobile genetic elements of the human gastrointestinal tract: potential for spread of antibiotic resistance genes. Gut Microbes. 2013 Jul-Aug;4(4):271-80. doi: 10.4161/gmic.24627. Epub 2013 Apr 12. PMID 23651955
- [Background] Fehily SR, Basnayake C, Wright EK, Kamm MA. Fecal microbiota transplantation therapy in Crohn's disease: Systematic review. J Gastroenterol Hepatol. 2021 Oct;36(10):2672-2686. doi: 10.1111/jgh.15598. Epub 2021 Jul 6. PMID 34169565
- [Background] Sokol H, Landman C, Seksik P, Berard L, Montil M, Nion-Larmurier I, Bourrier A, Le Gall G, Lalande V, De Rougemont A, Kirchgesner J, Daguenel A, Cachanado M, Rousseau A, Drouet E, Rosenzwajg M, Hagege H, Dray X, Klatzman D, Marteau P; Saint-Antoine IBD Network; Beaugerie L, Simon T. Fecal microbiota transplantation to maintain remission in Crohn's disease: a pilot randomized controlled study. Microbiome. 2020 Feb 3;8(1):12. doi: 10.1186/s40168-020-0792-5. PMID 32014035